CLINICAL TRIAL: NCT02364518
Title: TranQuill™ Sling Snoreplasty for Snoring and Mild Obstructive Sleep Apnea: A Single-arm, Pilot Study for Safety and Effectiveness
Brief Title: TranQuill™ Sling Snoreplasty for Snoring and Mild Obstructive Sleep Apnea:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TranQuill™ Sling Snoreplasty
Record Dates: First submitted 2014-04-15; First posted 2015-02-18 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Snoring; Obstructive Sleep Apnea
Keywords: Snoring; snoreplasy; Tranquill; Sutures
MeSH Terms: conditions — Snoring; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Snoreplasty (Experimental): Treatment of Snoring and/or mild obstructive sleep apnea with snoreplasty.
  Interventions: Procedure: Snoreplasty

INTERVENTIONS:
Procedure: Snoreplasty — The procedure will be performed under local anesthesia in the examination chair. The subject's throat will be anesthetized with benzocaine spray followed by infiltration of the soft palate with 4-5 milliliters of 1% lidocaine with 1:100,000 epinephrine. The TranQuill suture will be inserted into the soft palate tissues using a predescribed pattern.

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of TranQuillTM Sling (a suture or thread used in surgery that is knotless) in snoreplasty (surgery procedure) for the treatment of snoring and mild OSA in adult subjects. The TranQuill Sling Snoreplasty (QSS) is a procedure where the suture will be inserted into the soft palate tissues for the treatment of snoring and/or mild obstructive sleep apnea. Soft palate tissues are tissues in the back of the roof of the mouth.

The research results will be used to provide data on feasibility (strengths and weaknesses), safety, performance, and effectiveness data for the Surgical Specialties, Inc as a therapy for snoring and/or mild obstructive sleep apnea. The TranQuillTM Sling is approved by the U.S. Food and Drug Administration (FDA). The TranQuillTM Sling is used in all types of surgery that involved deep tissues in the body.

The investigator in charge of the study is Dr. Boyd Gillespie. MUSC and Dr. Gillespie receive financial support from Surgical Specialties, Inc. to conduct the study. MUSC is the only place that this study will be conducted. For this research study the investigators plan to enroll a total of up to 20 subjects at the Medical University of South Carolina.

DETAILED DESCRIPTION:
Study Methodology:

Subject Recruitment. Twenty subjects will be recruited from the MUSC Snoring Clinics as well as public information seminars held in the greater Charleston area. Attempts will be made to recruit both a gender and racially diverse study population.

Subject Screening. Subjects who are potentially eligible for the trial include patients who seek treatment chronic snoring disruptive to their bed-partner. Patients will require a pre-treatment assessment with a Watch-PAT home sleep study device to rule-out moderate and severe sleep apnea. Patients must have a regular bed-partner to participate in order to capture study outcomes.

Inclusion Criteria. Potential subjects must meet the following inclusion criteria:

* Age ≥ 22 years (no upper limit)
* Regular bed-partner
* Chronic, disruptive snoring according to bed-partner
* Snoring, upper airway resistance syndrome, or mild obstructive sleep apnea (AHI ≤ 15; lowest O2 saturation ≥ 85%) on home sleep testing with Watch-PAT
* No prior surgical treatment for snoring or OSAS other than nasal surgery
* Willing and capable of providing informed consent

Exclusion Criteria.

* Age < 22 years
* No regular bed-partner
* Intermittent or occasional snoring
* Moderate-to-severe obstructive sleep apnea (AHI ≥ 16; Lowest O2 sat <85%) or evidence of central apnea (≥ 10% of apneic events) on home sleep testing with Watch-PAT
* BMI ≥ 32 kg/m2
* Modified Mallampati 3 or 4
* Tonsil Grade 3 or 4
* Significant nasal obstruction (> 50% of nasal airway diameter on one side)
* Previous palatal surgery (cleft palate; uvulopalatopharyngoplasty; uvulectomy; Pillar implants; Somnoplasty)
* Current cigarette smoker (≥ 1 cigarette per day)
* Known history of coronary artery disease or stroke
* Chronic obstructive pulmonary disease (COPD)
* Diabetes
* Major depression or non-controlled psychiatric illness
* Drug or alcohol abuse
* Untreated or poorly controlled hypertension
* Anticoagulation therapy (ex. Coumadin or Plavix; single baby aspirin per day allowable)
* History of bleeding or clotting disorder
* Another significant sleep disorder (e.g., insomnia, periodic limb movement)
* Tonsillar hypertrophy
* Chronic Obstructive Pulmonary Disease (COPD)
* Interstitial Lung Disease (ILD)
* Cystic Fibrosis
* Acute Repiratory Distress Syndrome (ARDS)
* Nasal or supraglottic obstruction on fiberoptic examination
* ASA class III ,IV, V
* Latex allergy
* Lidocaine allergy
* Pregnancy or plans to become pregnant Note: women of childbearing potential must demonstrate a negative pregnancy test upon enrollment and/or be using an acceptable form of birth control (OCPs; IUD).
* Major depression or non-stabilized psychiatric disorder
* Drug or alcohol abuse
* Previous palatal or tongue surgery
* Stable or unstable angina
* CHF
* Moderate or severe valvular disease
* TIA/CVA
* Carotid stenosis or endarterectomy
* Anemia
* Room air SpO2 < 95%
* Pulmonary hypertension
* Dialysis
* Central or mixed apnea ≥ 10% of respiratory events
* Participation in another clinical study (enrolled in any concurrent study) whose investigational plan is judged to interfere or affect any of the measures of this study

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 22 years (no upper limit)
* Regular bed-partner
* Chronic, disruptive snoring according to bed-partner
* Snoring, upper airway resistance syndrome, or mild obstructive sleep apnea (AHI ≤ 15; lowest O2 saturation ≥ 85%) on home sleep testing with Watch-PAT
* No prior surgical treatment for snoring or OSAS other than nasal surgery
* Willing and capable of providing informed consent

Exclusion Criteria:

* Age < 22 years
* No regular bed-partner
* Intermittent or occasional snoring
* Moderate-to-severe obstructive sleep apnea (AHI ≥ 16; Lowest O2 sat <85%) or evidence of central apnea (≥ 10% of apneic events) on home sleep testing with Watch-PAT
* BMI ≥ 32 kg/m2
* Modified Mallampati 3 or 4
* Tonsil Grade 3 or 4
* Significant nasal obstruction (> 50% of nasal airway diameter on one side)
* Previous palatal surgery (cleft palate; uvulopalatopharyngoplasty; uvulectomy; Pillar implants; Somnoplasty)
* Current cigarette smoker (≥ 1 cigarette per day)
* Known history of coronary artery disease or stroke
* Chronic obstructive pulmonary disease (COPD)
* Diabetes
* Major depression or non-controlled psychiatric illness
* Drug or alcohol abuse
* Untreated or poorly controlled hypertension
* Anticoagulation therapy (ex. Coumadin or Plavix; single baby aspirin per day allowable)
* History of bleeding or clotting disorder
* Another significant sleep disorder (e.g., insomnia, periodic limb movement)
* Tonsillar hypertrophy
* Chronic Obstructive Pulmonary Disease (COPD)
* Interstitial Lung Disease (ILD)
* Cystic Fibrosis
* Acute Repiratory Distress Syndrome (ARDS)
* Nasal or supraglottic obstruction on fiberoptic examination
* ASA class III ,IV, V
* Latex allergy
* Lidocaine allergy
* Pregnancy or plans to become pregnant Note: women of childbearing potential must demonstrate a negative pregnancy test upon enrollment and/or be using an acceptable form of birth control (OCPs; IUD).
* Major depression or non-stabilized psychiatric disorder
* Drug or alcohol abuse
* Previous palatal or tongue surgery
* Stable or unstable angina
* CHF
* Moderate or severe valvular disease
* TIA/CVA
* Carotid stenosis or endarterectomy
* Anemia
* Room air SpO2 < 95%
* Pulmonary hypertension
* Dialysis
* Central or mixed apnea ≥ 10% of respiratory events
* Participation in another clinical study (enrolled in any concurrent study) whose investigational plan is judged to interfere or affect any of the measures of this study

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index | 90 days
  0-100
Oxygen Desaturation Index | 90 days
  0-100
Respiratory Disturbance Index | 90 days
  0-100
Bed Partner Scoring | 90 days
  0-10

CONTACTS AND LOCATIONS:
Overall Officials: M. Boyd Gillespie, MD, Principal Investigator — Medical University of South Carolina; Shaun A Nguyen, MD, MA, CPI, Principal Investigator — Medical University of South Carolina
Locations (1):
- Department of Otolaryngology- Head and Neck Surgery- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Murphey AW, Nguyen SA, Fuller C, Weber AC, Camilon MP, Gillespie MB. TranQuill sling snoreplasty for snoring: A single-arm pilot study for safety and effectiveness. Laryngoscope. 2016 Jan;126(1):243-8. doi: 10.1002/lary.25361. Epub 2015 Nov 4. PMID 26536156